CLINICAL TRIAL: NCT06709222
Title: Investigation of the Effectiveness of Dual-Task Exercises Applied in Addition to Robotic Rehabilitation in Hemiplegic Patients: A Randomized Controlled Trial
Brief Title: Robotic Rehabilitation and Dual-Task Exercises in Hemiplegic Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar17
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Coping; Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): the group that received robotic rehabilitation only
  Interventions: Other: robotic rehabilitation
- exercise (Experimental): group receiving robotic rehabilitation and dual-task exercises
  Interventions: Other: robotic rehabilitation; Other: exercise

INTERVENTIONS:
Other: robotic rehabilitation — robotic rehabilitation
Other: exercise — dual-task exercises
  Arms: exercise

SUMMARY:
The aim of this study was to investigate the effectiveness of dual-task exercises combined with robotic rehabilitation applied to post-stroke hemiplegia patients.

DETAILED DESCRIPTION:
This research is designed as a randomized controlled experimental study. The study will be conducted on 40 hemiplegic patients. Participants will be randomly divided into two groups. Patients in the exercise group will be subjected to dual-task exercises together with robotic rehabilitation. Patients in the control group will be subjected to only the robotic rehabilitation treatment program. Both groups will be treated with 30-45 minute sessions, 3 days a week for 6 weeks. The exercises will be explained to the patients in detail one-on-one and repeated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of post-stroke hemiplegia (hemiplegia onset must be between 3 months and 1 year).
* Age range: 30-60 years.
* Voluntariness to participate in rehabilitation.
* Patients with a motor function loss of 30-70% according to Fugl-Meyer Motor Assessment results.
* Literacy

Exclusion Criteria:

* History of active psychiatric disease.
* Severe joint deformities or other neurological diseases.
* Having had a recent stroke during rehabilitation.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-13 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Timed up and go test | 14 weeks
  Timed up and go test is used for the assessment of falls risk among elderly population. The Timed "Up and Go" (TUG) Test measures, in seconds, the time taken by an individual to stand up from a standard arm chair (approximate seat height of 46 cm, arm height 65 cm), walk a distance of 3 meters (approximately 10 feet), turn, walk back to the chair, and sit down.
  Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more.
  Clinical guide: <10 seconds = normal <20 seconds = good mobility, can go out alone, mobile without a gait aid <30 seconds = problems, cannot go outside alone, requires a gait aid A score of more than or equal to 14 seconds has been shown to indicate high risk of falls.
Improvement on Montreal Cognitive Assessment test of 5 points or more than baseline( total score is out of 30 points) | 14 weeks
  Subject will complete 3 Montreal Cognitive assessment prior to study over 1 week time. Best score of three is used.
  After study is complete subject will also undergo 3 Montreal cognitive assessment over 1 week immediately after study. Again best score is used.
Mini-Mental State Examination | 14 weeks
  Mini-Mental State Examination, 1 point for each correct answer maximun score: 30 - minimum score:24

CONTACTS AND LOCATIONS:
Overall Officials: Kübra UZUN, Study Chair — Uskudar University
Locations (1):
- Sancak Medical Center, Istanbul, Sancaktepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li Y, Lian Y, Chen X, Zhang H, Xu G, Duan H, Xie X, Li Z. Effect of task-oriented training assisted by force feedback hand rehabilitation robot on finger grasping function in stroke patients with hemiplegia: a randomised controlled trial. J Neuroeng Rehabil. 2024 May 14;21(1):77. doi: 10.1186/s12984-024-01372-3. PMID 38745227
- [Background] Ye JY, Chen R, Chu H, Lin HC, Liu D, Jen HJ, Banda KJ, Kustanti CY, Chou KR. Dual-task training in older adults with cognitive impairment: A meta-analysis and trial sequential analysis of randomized controlled trials. Int J Nurs Stud. 2024 Jul;155:104776. doi: 10.1016/j.ijnurstu.2024.104776. Epub 2024 Apr 18. PMID 38703695
- [Background] Uysal I, Ozden F, Tumturk I, Imerci A. The effectiveness of dual task exercise training on balance, mobility, physical performance, and quality of life in children with cerebral palsy: a single-blind randomized controlled trial. Ir J Med Sci. 2024 Apr;193(2):813-821. doi: 10.1007/s11845-023-03530-3. Epub 2023 Sep 30. PMID 37777679